CLINICAL TRIAL: NCT05344326
Title: Development and Piloting of a Low Intensity Cognitive Analytic-Informed Guided Self-help for Depression to be Used Within Increasing Access to Psychological Therapies (IAPT)
Brief Title: Cognitive Analytic-Informed Guided Self-help for Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 175377
Record Dates: First submitted 2022-01-12; First posted 2022-04-25 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Mixed methods, small N, case series
Masking Description: The PWP and service users will be aware of the intervention
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAT-GSH (Experimental): Participants, who provide informed consent, will be provided an assessment session, six fortnightly CAT-GSH sessions, and one follow-up session.
  Interventions: Other: Cognitive Analytic Therapy - Guided Self Help (CAT-GSH)

INTERVENTIONS:
Other: Cognitive Analytic Therapy - Guided Self Help (CAT-GSH) — CAT-GSH is a novel intervention designed to help those with depression by focusing on the relationships within their life. GSH is used in step two of IAPT services and is typically six fortnightly sessions where the PWP helps the service user complete the self help manual.

SUMMARY:
Cognitive analytic therapy (CAT) is used within mental health services as a treatment for a range of mental health difficulties. Recent research has adapted CAT to be used as guided self-help for anxiety within Increasing Access to Psychological Therapies (IAPT). IAPT is a mental health service. Guided self help-CAT (CAT-GSH) is delivered by mental health professionals called Psychological Wellbeing Practitioners (PWPs). This current study aims to develop and pilot a CAT-GSH manual for depression for use in the same context and practitioners. Stage one uses past research and consultation meetings to help develop the treatment. Stage two will use different approaches to explore the acceptability and outcomes of the intervention.

DETAILED DESCRIPTION:
Aims Phase One

1) Develop a CAT-informed GSH manual (CAT-GSH) for depression Phase Two

1. Pilot CAT-SH within IAPT setting
2. To explore the impact of CAT-GSH on outcomes
3. To investigate the acceptability of CAT-GSH

Method Stage One Past research and consultation meetings will be consolidated into a matrix. This will inform the development of the treatment manual.

Stage Two A mixed-methods, small N case series design will be utilized to pilot the CAT-GSH manual within IAPT services. Three Psychological Wellbeing Practitioners (PWP) and 10 service users will be recruited from Barnsley IAPT service. The PWPs will be provided a two-day training course before the study begins. This will cover information regarding the CAT-GSH, data management, and the protocol. To recruit 10 service user participants, it is predicted the first 60 people on the Barnsley IAPT waiting list would need to be screened to account for eligibility criteria, preference, and attrition.

Participants will be offered to complete CAT-GSH if:

1. Depression is the main problem
2. They score above the clinical cut off (10 points) on the Patient Health Questionnaire (PHQ9; Kroenke and Spitzer, 2002)
3. Aged between 18 - 65
4. Would prefer to use CAT-GSH over other interventions
5. Consent to participate in study
6. Can engage with reading materials

The exclusion criteria will be:

1. Patients who would normally be 'stepped up' due to complexity and risk
2. Patients are receiving other therapies
3. Substance users unable to abstain during sessions The exclusion criteria are in line with IAPT step-two treatment guidance and support.

The participants will be invited to an assessment session where they will be informed about the research, be provided with information sheets and consent sheets. The participants will have time to contact the researchers if they have any questions about the research.

If they provide informed consent, they will be provided with six, fortnightly CAT-GSH sessions facilitated by the PWPs. In these sessions, they will also complete three outcome measures. The patient health questionnaire, the generalized anxiety disorder assessment, and the work and social adjustment scale.

They will receive a follow-up session, with the PWP, where they will also complete the outcome measures and review their care. They will also arrange an interview with the primary research to explore their experiences of CAT-GSH. This will follow an interview schedule. The PWPs will also attend a separate, PWP group interview where they will also reflect on their experiences of delivering GSH. This will be provided by the researcher.

The analysis stage of the process will then begin as the researchers explore the outcome measure data and the interview data.

ELIGIBILITY:
Inclusion Criteria:

* Depression is the main problem
* They score above the clinical cut off (10 points) on the Patient Health Questionnaire (PHQ9; Kroenke and Spitzer, 2002)
* Aged between 18 - 65
* Would prefer to use CAT-GSH over other interventions
* Consent to participate in study
* Can engage with reading materials

Exclusion Criteria:

* Patients who would normally be 'stepped up' due to complexity and risk
* Patients are receiving other therapies
* Substance users unable to abstain during sessions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2022-11-07 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Patient Health Questionnaire - PHQ9 | Through participant involvement, roughly 4 months. Administered 8 times across assessment, treatment, and follow up. Once during assessment, weekly during intervention (6 times). Follow-up outcomes will be collected between 4-8 weeks after intervention.
  The PHQ9 is a 9-item self-administered questionnaire designed for detecting depression and is based on the DSM-IV criteria.
Generalised Anxiety Disorder Assessment - GAD 7 | Through participant involvement, roughly 4 months. Administered 8 times across assessment, treatment, and follow up. Once during assessment, weekly during intervention (6 times). Follow-up outcomes will be collected between 4-8 weeks after intervention.
  The GAD7 is also widely used within primary care settings and is a self-reported screening tool for generalised anxiety disorder.
Work and Social Adjustment Scale - WSAS | Through participant involvement, roughly 4 months. Administered 8 times across assessment, treatment, and follow up. Once during assessment, weekly during intervention (6 times). Follow-up outcomes will be collected between 4-8 weeks after intervention.
  This scale measures social functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kelly, Principal Investigator — University of Sheffield
Locations (1):
- Barnsley IAPT Service, Barnsley, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Only anonymized data will be shared. Personal data will not be.
Supporting Information: Study Protocol
Time Frame: At the end of the study (approximately May 2023), data will be stored on the University of Sheffield's ORDA (online research hub) for 5 years according to the University of Sheffield's retention period.
Access Criteria: Information can be requested through ORDA by those who qualify for membership.